CLINICAL TRIAL: NCT00867568
Title: A Phase 1 Trial of TPI 287 as a Single Agent and in Combination With Temozolomide in Patients With Refractory or Recurrent Neuroblastoma or Medulloblastoma
Brief Title: TPI 287 in Patients With Refractory or Recurrent Neuroblastoma or Medulloblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI-287
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma; Medulloblastoma; Relapse
Keywords: Relapsed Neuroblastoma; Refractory Neuroblastoma; Relapsed Medulloblastoma; Refractory Medulloblastoma
MeSH Terms: conditions — Neuroblastoma; Medulloblastoma; Recurrence | interventions — TPI-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TPI 287 (Experimental)
  Interventions: Drug: TPI 287

INTERVENTIONS:
Drug: TPI 287 — Three patients will be enrolled to receive single agent TPI 287 IV administered on Days 1, 8 and 15 of the first and second 28-day cycle. The starting dose of 90 mg/m2 (Dose Level 1) is 75% of the established adult MTD for this schedule in adults, which is 125 mg/m2. Dose escalation will take place in a standard 3+3 design, in which doses will increase by approximately 20 to 25% in successive 3-patient cohorts.

SUMMARY:
The purpose of this research study is to evaluate a new investigational drug (TPI 287) for neuroblastoma and medulloblastoma both alone and in combination with temozolomide (a currently approved drug). An investigational drug is one that has not yet been approved by the Food and Drug Administration. This investigational drug is called TPI 287. This study will look at the safety and tolerability of TPI 287 both alone and in combination with temozolomide, and look to establish a safe dose of this agent. The study will also look at the tumor's response to these drugs, but this is not the primary objective of this study.

TPI 287 was shown to be effective in stopping tumor growth and was also shown to be safe in three different animal species. TPI 287 has been tested in humans in four clinical trials, and approximately 100 subjects with various types of cancers have received the drug. All of these subjects that have received TPI 287 have been adults. TPI 287 has not been tested in a pediatric population before this study.

Temozolomide was tested in recurrent neuroblastoma and showed activity in a recently published study. Preclinical studies of TPI in combination with temozolomide have shown at minimum an additive effect. The ability of temozolomide and TPI 287 to be effective in combination is suggested by these two drugs showing even greater activity when used together.

DETAILED DESCRIPTION:
Neuroblastoma:

Neuroblastoma is the most common pediatric extracranial solid tumor and accounts for 7% to 10% of childhood cancers (American Cancer Society 2008; Bernstein et al. 1992). Whereas the prognosis for infants with neuroblastoma is generally good, currently only 30% of children diagnosed after 12-15 months of age survive despite aggressive multimodal therapies (Brodeur et al 1993; Park et al 2008). High-dose chemotherapy (HDC) followed by hematopoietic stem cell transplantation (HSCT) and maintenance therapy with retinoic acid improves survival by 35% in children presenting with metastatic NB, but the 5-year event-free survival remains below 50% (Matthay et al, 1999; Hartmann, et al, 1999). Consequently, the evaluation of new drugs is strongly needed in this disease.

1.2

Medulloblastoma:

Medulloblastoma is the most common malignant brain tumor in children and accounts for 16% of all brain tumors in children 0-14 years old and 6% in adolescents 15-19 years old (CBTRUS 2008). Current therapies for children with disseminated disease are associated with severe long-term toxicities, and lead to cure in only a minority of cases. (Partap et al, 2007). Thus, the development of new therapies-especially ones with more favorable toxicity profiles-would represent a significant improvement in the treatment of this disease. Although there have been reports that the survival rate of children with chemosensitive relapsed medulloblastoma can approach 40% following intensive chemotherapy combined with autologous stem cell support, more recent data looking at survival of all patients relapsing after modern combination chemotherapy and radiation is also on the order of 10-15%. (Rood, et al, 2004) As such, new therapeutic approaches are needed to treat these children.

1.3 The Investigational Product TPI 287 1.3.1

Preclinical Studies:

Tapestry Pharmaceuticals, Inc. developed a novel anti-microtubule agent, TPI 287, for which Archer Biosciences, Inc. is now the sponsor. TPI 287 is synthetically manufactured from naturally occurring taxanes extracted from yew starting material. The synthesis involves modifications of the side chain to make the drug more lipophilic, and modification of the baccatin ring structure with the intent of circumventing MDR-based resistance and allowing for binding to mutant tubulin. Selection of TPI 287 was also made on the basis of the very high potency of this drug against several neuroblastoma cell lines and xenograft models (see below).

In vitro, TPI 287 was shown to have comparable cytotoxicity to paclitaxel in several MDR- cell lines, but was 5 - 3900-fold more active than several comparator compounds in MDR+ cells lines. In MCF-7-AR breast cancer cells, which display MDR-based resistance, TPI 287 was 20-times more active than paclitaxel. Similar findings were observed in MDR+ cells derived from colorectal, breast and prostate cancers, as well as from neuroblastoma, as noted.TPI 287 was also evaluated in a variety of xenograft models. As in vitro, TPI 287 was superior to paclitaxel in vivo in the MCF-7-AR xenograft. TPI 287 also had superior activity when compared to SN-38 in the HCT-15 and HCT-116 colon cancer xenografts; when compared to docetaxel in the PC3 prostate cancer xenograft; and when compared to docetaxel and doxorubicin in the MV522 NSCLC xenograft.

Activity against glioblastoma was shown in transplanted xenografts, and efficacy was demonstrable using both IV and oral administration. In addition, in an orthotopic xenograft using U251 cells implanted in the brains of nude mice, treatment with either TPI 287, temozolomide, or combinations were compared to control animals, evaluating median survival (10 animals per group) as well as animals whose survival extended beyond 110 days. The results of this study, repeated for corroboration at an outside facility, are shown in Table 4. Significant synergy and improvement in long term survival can be seen with the combination of temozolomide (TMZ) plus TPI 287.Potent activity had also been shown against neuroblastoma cell lines as previously noted, and this was also demonstratable in transplanted xenografts, showing greater activity than paclitaxel, docetaxel or nab-paclitaxel. Studies recently completed (Sholler, et al, personal communication) show TPI 287 has activity against additional neuroblastoma cell lines as well as medulloblastoma cell lines and increased efficacy when TPI 287 is combined with TMZ in neuroblastoma.Toxicology studies demonstrated that TPI 287 was generally well tolerated. The MTD in the rat was 48 mg/kg and in the dog, 12.5 mg/kg. Toxicity was primarily characterized by bone marrow suppression and mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven neuroblastoma and confirmation of refractory or recurrent disease or medulloblastoma with histologic confirmation at diagnosis or at the time of recurrence/progression
* Patients must be age >12 months and diagnosed before the age of 21
* Life expectancy must be more than 3 months
* If measurable disease, this must be demonstrated by residual abnormal tissue at a primary or metastatic site measuring more than 1 cm in any dimension by standardized imaging (CT or MRI). For patients with neuroblastoma who only have skeletal disease, there must be at least two persisting skeletal foci on meta-iodobenzylguanidine (MIBG) follow-up scans
* Current disease state must be one for which there is currently no known curative therapy
* Lansky Play Score must be more than 30 and/or ECOG performance status must be 0 to 2
* For patients with medulloblastoma receiving steroids, the dose must be stable (i.e. not increasing) for at least one week before starting study
* Patients without bone marrow metastases must have an ANC > 750/μl and platelet count >50,000/μl
* Adequate liver function must be demonstrated, defined as:

  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND
  * SGPT (ALT) < 10 x upper limit of normal (ULN) for age
* No other significant organ toxicity defined as > Grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events version 3 (NCI-CTCAE V3.0 (http://ctep.cancer.gov/forms/CTCAEv3.pdf))
* A negative urine pregnancy test is required for female participants of child bearing potential (≥13 years of age or after the onset of menses)
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these can not be used, contraceptive foam with a condom is recommended
* Informed Consent: All patients and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines
* Patients may have received microtubulin inhibitors and/or temozolomide during previous therapies

Exclusion Criteria:

* Patients who have received any chemotherapy administered within the last 21 days
* Patients who have received radiotherapy within the last 30 days
* Patients who have received myeloablative therapy within the previous 3 months
* Patients receiving anti-tumor therapy for their disease or any investigational drug concurrently
* Patients with serious infection or a life-threatening illness (unrelated to tumor) that is > Grade 2 (NCI CTCAE V3.0), or active, serious infections requiring parenteral antibiotic therapy within 4 weeks prior to screening
* Any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a patient's ability to sign or the legal guardian's ability to sign the informed consent, and patient's ability to cooperate and participate in the study
* Patients with known hypersensitivity to any of the components of the drugs to be administered on study
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (6):
- United States (6):
  - Rady Children's Hospital, San Diego, California
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - UVM/FAHC, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Beat Childhood Cancer — https://beatcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TPI 287
Started | 18
Completed | 3
Not Completed | 15
Not completed — Lack of Efficacy | 10
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TPI 287
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] — One subject, age 25, was allowed to enroll on study, but was censored from endpoints due to age.
  years | 7.5 [4 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: To determine the safety, tolerability and maximum tolerated dose (MTD) of TPI 287 as a single agent and collect exploratory data on the safety and tolerability of TPI 287 in combination with temozolomide (TMZ) in pediatric and young adult patients with refractory or recurrent neuroblastoma or medulloblastoma
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | TPI 287
Number analyzed (Participants) | 18
participants | 14

2. Secondary Outcome: Tmax of TPI 287in Pediatrics Using Pharmacokinetic (PK) Testing.
Time Frame: Cycle 3 day 1 at Pre dose, 0 (end of infusion), 0.25, 0.5, 1, 2, 4, and 6 hours post dose
Population: Six patients at the MTD dose of 125mg/m2/dose
Measure: Mean (Full Range); unit: hour
Arm/Group | TPI 287
Number analyzed (Participants) | 6
hour | 1 [1 to 1]

3. Secondary Outcome: Number of Patients With an Overall Response Rate (ORR) of PR or CR
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: 18 subjects enrolled, one subject censored due to age, 5 subjects not evaluable. Analysis population= 12 patients.
Measure: Number; unit: participants
Arm/Group | TPI 287
Number analyzed (Participants) | 12
participants | 1

4. Secondary Outcome: Progression Free Survival (PFS) of Participants Using Days From Start of Study Drug Until Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 4 years
Population: 18 subjects enrolled, one subject censored due to age, 5 subjects not evaluable. Analysis population= 12 patients.
Measure: Mean (Full Range); unit: months
Arm/Group | TPI 287
Number analyzed (Participants) | 12
months | 6.2 [0.4 to 36.4]

5. Secondary Outcome: Cmax of TPI 287in Pediatrics Using Pharmacokinetic (PK) Testing.
Time Frame: Cycle 3 day 1 at Pre dose, 0 (end of infusion), 0.25, 0.5, 1, 2, 4, and 6 hours post dose
Population: Six patients at the MTD dose of 125mg/m2/dose
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | TPI 287
Number analyzed (Participants) | 6
ng/ml | 3435.00 (872.61)

6. Secondary Outcome: AUC of TPI 287in Pediatrics Using Pharmacokinetic (PK) Testing.
Time Frame: Cycle 3 day 1 at Pre dose, 0 (end of infusion), 0.25, 0.5, 1, 2, 4, and 6 hours post dose
Population: Six patients at the MTD dose of 125mg/m2/dose
Measure: Mean (Standard Error); unit: ng*hr/mL
Arm/Group | TPI 287
Number analyzed (Participants) | 6
ng*hr/mL | 5474.90 (684.96)

ADVERSE EVENTS:
Time Frame: New adverse events collected from first dose of study drug to 30 days past last dose of study drug. Related adverse events followed until resolution, approximately 1 year.
Arm/Group | TPI 287
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 (N=18)
Seizure (Nervous system disorders) | 1 (1) — Seizure related to disease in CNS, not related to study drug.
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1)
Progression of disease resulting in death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 (N=18)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Albumin Increase (Blood and lymphatic system disorders) | 1 (1)
ALT increase (Hepatobiliary disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)
AST Increase (Hepatobiliary disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Drug Reaction (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
GGT Increase (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
INR (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Rash- Lip sore (Skin and subcutaneous tissue disorders) | 1 (1)
Liver dysfunction (Hepatobiliary disorders) | 1 (1)
Neuropathic pain (Nervous system disorders) | 1 (1)
Neuropathy sensory (Nervous system disorders) | 2 (2)
Pain (General disorders) | 4 (4)
Seizure (Nervous system disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
SIADH (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less